CLINICAL TRIAL: NCT02831842
Title: A Non-Interventional Multi-country Study to Evaluate the Real World Effectiveness of Avastin (Bevacizumab) for First Line Treatment of Patients With Metastatic Colorectal Cancer and Known KRAS Status
Brief Title: A Real World Study to Evaluate Effectiveness of Avastin (Bevacizumab) for First Line Treatment of Patients With Metastatic Colorectal Cancer and Known KRAS Status
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MO30177
Record Dates: First submitted 2016-07-12; First posted 2016-07-13 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- mCRC Participants: Data of mCRC participants who received first-line treatment with bevacizumab-containing regimen or with chemotherapy alone and had KRAS-mutant status and mCRC participants who received first-line treatment with bevacizumab-containing regimen or an anti-epidermal growth factor receptor (EGFR)-containing regimen and had KRAS wild type status, will be collected retrospectively.
  Interventions: Drug: Anti-EGFR-Containing Regimen; Drug: Bevacizumab-containing regimen; Drug: Chemotherapy

INTERVENTIONS:
Drug: Anti-EGFR-Containing Regimen — Study protocol does not specify any particular chemotherapy regimen. The data will be collected retrospectively.
Drug: Bevacizumab-containing regimen — Study protocol does not specify any particular bevacizumab containing regimen. The data will be collected retrospectively.
  Other Names: Avastin
Drug: Chemotherapy — Study protocol does not specify any particular chemotherapy regimen. The data will be collected retrospectively.

SUMMARY:
This non-interventional study will meta-analyze overall survival outcomes among the participants with metastatic colorectal cancer (mCRC) with available V-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) status, who received firstline treatment with bevacizumab containing treatment regimen in routine clinical practice. The study leveraging secondary data from existing cohorts in the United Stats of America (USA), Germany, Australia, and Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Participants with metstatic colorectal cancer (mCRC) diagnosed at any point prior to March 2014 (United States [US] - Vector Oncology Protocol Sponsored by US Roche Pharma Medical Affairs), diagnosed between September 2006 and March 2015 (Germany - Tumourregister Kolorektales Karzinom [TKK] Registry Study Supported by German Roche Pharma Affiliate), diagnosed between September 2009 and December 2014 (Australia - Treatment of Recurrent and Advanced Colorectal Cancer [TRACC] Registry Supported by Roche Pharma Australia), diagnosed between 2009 and 2013 (Denmark - Roche Diagnostic Sponsored Study and Aarhus University Hospital, Department of Clinical Epidemiology)
* Participants have been treated in first line with bevacizumab or Anti-EGFR treatment regimen or chemotherapy alone
* Participants have to have available data on overall survival (OS), KRAS testing status, and left/right tumor location status

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with mCRC and known KRAS status who received bevacizumab as first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 4278 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2016-06-09 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) in Participants With mCRC and a Documented KRAS Mutation who Received Bevacizumab-Containing Treatment or Chemotherapy Alone in Routine Clinical Practice | start of first-line therapy to death from any cause, or to last date known that participant is alive (retrospective data collection over approximately 9 years)

SECONDARY OUTCOMES:
OS in Participants With mCRC and a Documented KRAS Wild Type Status who Received Bevacizumab-Containing Treatment or Anti-EGFR Treatment in Routine Clinical Practice | start of first-line therapy to death from any cause, or to last date known that participant is alive (retrospective data collection over approximately 9 years)

CONTACTS AND LOCATIONS:
Overall Officials: Germany: PEI Clinical Trials, Study Director — Hoffmann-La Roche